CLINICAL TRIAL: NCT00904670
Title: NWP06 in the Treatment of Children With Attention Deficit Hyperactivity Disorder (ADHD)- A Laboratory Classroom Study
Brief Title: Quillivant Oral Suspension (Quillivant XR) in the Treatment of Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NWP06-ADD-100; B7491007
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-05

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Hyperactivity Attention Deficit Disorder; ADHD; Pediatric Patients; Quillivant; methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: Quillivant Oral Suspension XR; Drug: Placebo
- Comparator (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quillivant Oral Suspension XR — Oral Suspension 25mg/5mL; 20-60 mg/day
  Other Names: methylphenidate hydrochloride oral suspension
  Arms: Active
Drug: Placebo — Matching Placebo Oral Suspension 25mg/5mL; 20-60 mg/day
  Arms: Active
Drug: Placebo — Matching placebo was a solution that was identical in taste and appearance to the Active drug that was used in this study.
  Arms: Comparator

SUMMARY:
The objective of this study was to establish that an optimal dose of Quillivant XR oral suspension would result in a significant reduction in signs and symptoms of ADHD compared to placebo treatment in pediatric patients ages 6-12 years with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female from 6 to 12 years of age at the time of screening, inclusive.
* Diagnosis of ADHD by a Psychiatrist, Psychologist, Developmental Pediatrician, or a Pediatrician meeting diagnostic criteria for ADHD (DSM-IV). A Schedule for Affective Disorders and Schizophrenia for School Age Children (K-SADS)16 was administered on all subjects to assist in diagnostic process.
* A clinician-administered Clinical Global Impression of Severity (CGI-S) score of 3 or greater. An Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS) score at screening or baseline greater than or equal to the 90th percentile normative values for gender and age in at least one of the following categories: the hyperactive-impulsive subscale, inattentive subscale or the total score.
* Subject must have been in need of pharmacological treatment for ADHD.
* Subjects taking a medication to control ADHD at the time of screening must have been experiencing suboptimal efficacy, a safety or tolerability issue or in need of a long-acting liquid formulation.
* For subjects taking any daily medication at screening aside from ADHD medication: parent or legal guardian agreed that there would be no elective changes in subject's medications during the study (10 weeks total).

Exclusion Criteria:

* Excluded comorbid psychiatric diagnoses: DSM-IV Axis I diagnosis (active) other than ADHD, with the exception of Specific Phobias, Learning Disorders, Motor Skills Disorders, Communication Disorders, Oppositional Defiant Disorder, Elimination Disorders, Sleep Disorders, and Adjustment Disorders.
* Clinically significant cognitive impairment as assessed in the clinical judgment of the Investigator. In cases where this was not clear, study staff were permitted to administer a Wechsler Abbreviated Scale of Intelligence (WASI)17 to estimate the intelligence quotient (IQ). Significant cognitive impairment for this protocol was defined as an estimated IQ below 80.
* Subjects with chronic medical illnesses including seizure disorder (excluding a history of febrile seizures), severe hypertension, thyroid disease, structural cardiac disorders, serious cardiac conditions, serious arrhythmias, cardiomyopathy, glaucoma, Tourette's Disorder, family history of Tourette's Disorder or tics.
* Use of monoamine oxidase inhibitors within 30 days of the screening visit.
* Use of any psychotropic medication (except sedative hypnotics prescribed as a sleep aid at a stable dose for at least 30 days prior to screening, at bedtime only). Use of stimulant medication for control of ADHD at screening was permitted if inclusion criterion number 6 was met.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - UC Irvine Child Development Center, Irvine, California
  - Center for Psychiatry and Behavioral Medicine, Incorporated, Las Vegas, Nevada

REFERENCES:
- [Derived] Wigal SB, Childress AC, Belden HW, Berry SA. NWP06, an extended-release oral suspension of methylphenidate, improved attention-deficit/hyperactivity disorder symptoms compared with placebo in a laboratory classroom study. J Child Adolesc Psychopharmacol. 2013 Feb;23(1):3-10. doi: 10.1089/cap.2012.0073. Epub 2013 Jan 5. PMID 23289899
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=NWP06-ADD-100&StudyName=Quillivant%20Oral%20Suspension%20%28Quillivant%20XR%29%20in%20the%20Treatment%20of%20Attention%20Deficit%20Hyperactivity%20Disorder%20%28ADHD%29

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of an open-label (OL) dose-optimization phase (4 to 6 weeks), and a placebo-controlled, double blind (DB) 2-way crossover phase (1 week each) with no dose adjustments.
Groups:
- OL Phase (NWP06); DB Phase (Placebo First, Then NWP06): Placebo-matched to NWP06 oral suspension once daily for 1 week in the first intervention period followed by NWP06 oral suspension at a once daily optimized dose (optimized during the 4 to 6 weeks open label phase at a starting dose of 20 milligram [mg] and titrated at a 10 or 20 mg increments, based on clinical response and tolerability to a maximum daily dose of 60 mg/day) for 1 week in the second intervention period.
- OL Phase (NWP06); DB Phase (NWP06 First, Then Placebo): NWP06 oral suspension at a once daily optimized dose (optimized during the 4 to 6 weeks open label phase at a starting dose of 20 milligram [mg] and titrated at a 10 or 20 mg increments, based on clinical response and tolerability to a maximum daily dose of 60 mg/day) for 1 week in the first intervention period followed by placebo-matched to NWP06 oral suspension once daily for 1 week in the second intervention period.
Period: Open Label Phase
Arm/Group | OL Phase (NWP06); DB Phase (Placebo First, Then NWP06) | OL Phase (NWP06); DB Phase (NWP06 First, Then Placebo)
Started | 23 | 22
Completed | 17 | 22
Not Completed | 6 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: First Intervention Period
Arm/Group | OL Phase (NWP06); DB Phase (Placebo First, Then NWP06) | OL Phase (NWP06); DB Phase (NWP06 First, Then Placebo)
Started | 17 | 22
Completed | 17 | 22
Not Completed | 0 | 0
Period: Second Intervention Period
Arm/Group | OL Phase (NWP06); DB Phase (Placebo First, Then NWP06) | OL Phase (NWP06); DB Phase (NWP06 First, Then Placebo)
Started | 17 | 22
Completed | 17 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 dose of study medication (either NWP06 or matching placebo) with at least 1 post-baseline safety assessment.
Groups:
- Entire Study Population: Includes all randomized participants who received at least 1 dose of study medication.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.8 (1.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 33

OUTCOME MEASURES:

1. Primary Outcome: Swanson, Kotin, Agler, M-Flynn, and Pelham Rating Scale (SKAMP)-Combined Scores at Hour 4 Post-Dose
Description: The SKAMP scale measures the manifestations of attention deficit hyperactivity disorder (ADHD) using an independent observer rating of the participant's impairment in classroom observed behaviors. SKAMP combined score is comprised of 13 items (including subscales: attention with items 1-4, deportment with items 5-8, quality of work with items 9-11 and compliance with items 12-13). The SKAMP composite score was obtained by summing up each item score where each item is rated on a 7-point impairment scale (0=normal to 6=maximal impairment) for a total possible combined score of 0 to 78; where higher score signified worst impairment.
Time Frame: Hour 4 post-dose
Population: Intent-to-Treat (ITT) analysis set included all randomized participants who received at least 1 dose of study medication (either NWP06 or matching placebo) and had at least 1 post-baseline efficacy assessment. N (number of participants analyzed)= participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- NWP06: NWP06 oral suspension at a once daily optimized dose (optimized during the 4 to 6 weeks open label phase at a starting dose of 20 milligram [mg] and titrated at a 10 or 20 mg increments, based on clinical response and tolerability to a maximum daily dose of 60 mg/day) for 1 week in either of the 2 intervention periods.
- Placebo: Placebo-matched to NWP06 oral suspension once daily for 1 week in either of the 2 intervention periods.
Arm/Group | NWP06 | Placebo
Number analyzed (Participants) | 39 | 39
units on a scale | 7.1 (5.64) | 19.3 (8.38)
Statistical Analysis 1: Comparison: NWP06 vs Placebo; Treatment comparisons for observed scores were assessed using linear models with sequence (Placebo/NWP06 and NWP06/Placebo), period, and treatment (NWP06 and Placebo) as fixed effects, and participant within sequence as a repeated effect with a compound symmetry correlation structure. A negative point difference indicated a positive effect of NWP06 over Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA; Least Square (LS) mean difference = -12.46, 95% CI 2-sided [-14.75 to -10.17], Standard Error of Mean 1.13

2. Secondary Outcome: Onset and Duration of Clinical Effect Based on SKAMP-Combined Scale
Description: Onset and duration is determined using SKAMP combined rating scale at each post-dose time point. Onset of effect is defined as first assessment time showing statistical significance (i.e. p is less than or equal to [=<] 0.05) between NWP06 and placebo and duration of effect is defined as the as last consecutive time-point at which difference is still statistically significant between NWP06 and placebo. SKAMP scale measures the manifestations of ADHD using an independent observer rating of the participant's impairment in classroom observed behaviors. SKAMP combined score is comprised of 13 items [subscales: attention (1-4 items), deportment (5-8 items), quality of work (9-11 items) and compliance (12-13 items)]. SKAMP combined score is obtained by summing up each item score where each item is rated on a 7-point impairment scale (0=normal to 6=maximal impairment) for total possible combined score of 0 to 78; where higher score signified worst impairment.
Time Frame: 0.75, 2, 8, 10, 12 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NWP06 | Placebo
Number analyzed (Participants) | 39 | 39
units on a scale
  Hour 0.75 | 9.5 (5.77) | 15.8 (7.25)
  Hour 2 | 7.2 (4.73) | 16.9 (7.96)
  Hour 8 | 10.8 (8.23) | 20.0 (9.33)
  Hour 10 | 14.0 (9.50) | 17.7 (9.04)
  Hour 12 | 15.1 (9.38) | 19.8 (10.91)
Statistical Analysis 1: Comparison: NWP06 vs Placebo; Hour 0.75: Treatment comparisons for observed scores were assessed using linear models with sequence (Placebo/NWP06 and NWP06/Placebo), period, and treatment (NWP06 and Placebo) as fixed effects, and participant within sequence as a repeated effect with a compound symmetry correlation structure. A negative point difference indicated a positive effect of NWP06 over Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean difference = -6.32, 95% CI 2-sided [-8.53 to -4.11], Standard Error of Mean 1.09
Statistical Analysis 2: Comparison: NWP06 vs Placebo; Hour 2: Treatment comparisons for observed scores were assessed using linear models with sequence (Placebo/NWP06 and NWP06/Placebo), period, and treatment (NWP06 and Placebo) as fixed effects, and participant within sequence as a repeated effect with a compound symmetry correlation structure. A negative point difference indicated a positive effect of NWP06 over Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean difference = -9.98, 95% CI 2-sided [-12.04 to -7.91], Standard Error of Mean 1.02
Statistical Analysis 3: Comparison: NWP06 vs Placebo; Hour 8: Treatment comparisons for observed scores were assessed using linear models with sequence (Placebo/NWP06 and NWP06/Placebo), period, and treatment (NWP06 and Placebo) as fixed effects, and participant within sequence as a repeated effect with a compound symmetry correlation structure. A negative point difference indicated a positive effect of NWP06 over Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean difference = -9.33, 95% CI 2-sided [-11.92 to -6.75], Standard Error of Mean 1.28
Statistical Analysis 4: Comparison: NWP06 vs Placebo; Hour 10: Treatment comparisons for observed scores were assessed using linear models with sequence (Placebo/NWP06 and NWP06/Placebo), period, and treatment (NWP06 and Placebo) as fixed effects, and participant within sequence as a repeated effect with a compound symmetry correlation structure. A negative point difference indicated a positive effect of NWP06 over Placebo; Test type: Superiority or Other; p = 0.0016, ANOVA; LS mean difference = -3.79, 95% CI 2-sided [-6.04 to -1.54], Standard Error of Mean 1.11
Statistical Analysis 5: Comparison: NWP06 vs Placebo; Hour 12: Treatment comparisons for observed scores were assessed using linear models with sequence (Placebo/NWP06 and NWP06/Placebo), period, and treatment (NWP06 and Placebo) as fixed effects, and participant within sequence as a repeated effect with a compound symmetry correlation structure. A negative point difference indicated a positive effect of NWP06 over Placebo; Test type: Superiority or Other; p = 0.0016, ANOVA; LS mean difference = -4.77, 95% CI 2-sided [-7.61 to -1.94], Standard Error of Mean 1.40

3. Secondary Outcome: SKAMP Attention Subscale Score Over 12 Hours
Description: SKAMP scale measures the manifestations of ADHD using an independent observer rating of the participant's impairment in classroom observed behaviors. SKAMP combined score is comprised of 13 items [subscales: attention (1-4 items), deportment (5-8 items), quality of work (9-11 items) and compliance (12-13 items)]. SKAMP combined score is obtained by summing up each item score where each item is rated on a 7-point impairment scale (0=normal to 6=maximal impairment) for total possible combined score of 0 to 78; where higher score signified worst impairment. SKAMP attention subscale is reported which evaluates concentration in the classroom and comprises of 4 items, with a total possible score for of 0 to 24; higher score indicates worst impairment.
Time Frame: 0.75, 2, 4, 8, 10, 12 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NWP06 | Placebo
Number analyzed (Participants) | 39 | 39
units on a scale
  Hour 0.75 | 1.3 (1.64) | 2.5 (2.52)
  Hour 2 | 1.1 (1.85) | 2.6 (2.93)
  Hour 4 | 0.9 (1.97) | 3.1 (3.49)
  Hour 8 | 1.2 (1.96) | 2.7 (3.58)
  Hour 10 | 2.5 (2.80) | 3.0 (3.43)
  Hour 12 | 2.4 (2.66) | 3.4 (3.11)
Statistical Analysis 1: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0051, ANOVA; LS mean difference = -1.12, 95% CI 2-sided [-1.88 to -0.36], Standard Error of Mean 0.38
Statistical Analysis 2: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean difference = -1.59, 95% CI 2-sided [-2.23 to -0.95], Standard Error of Mean 0.31
Statistical Analysis 3: Comparison: NWP06 vs Placebo; Hour 4: Treatment comparisons for observed scores were assessed using linear models with sequence (Placebo/NWP06 and NWP06/Placebo), period, and treatment (NWP06 and Placebo) as fixed effects, and participant within sequence as a repeated effect with a compound symmetry correlation structure. A negative point difference indicated a positive effect of NWP06 over Placebo; Test type: Superiority or Other; p = 0.0001, ANOVA; LS mean difference = -2.28, 95% CI 2-sided [-3.37 to -1.20], Standard Error of Mean 0.54
Statistical Analysis 4: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0055, ANOVA; LS mean difference = -1.49, 95% CI 2-sided [-2.52 to -0.47], Standard Error of Mean 0.51
Statistical Analysis 5: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.1977, ANOVA; LS mean difference = -0.54, 95% CI 2-sided [-1.38 to 0.29], Standard Error of Mean 0.41
Statistical Analysis 6: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.0491, ANOVA; LS mean difference = -0.88, 95% CI 2-sided [-1.76 to 0.00], Standard Error of Mean 0.43

4. Secondary Outcome: SKAMP Deportment Subscale Score Over 12 Hours
Description: SKAMP scale measures the manifestations of ADHD using an independent observer rating of the participant's impairment in classroom observed behaviors. SKAMP combined score is comprised of 13 items [subscales: attention (1-4 items), deportment (5-8 items), quality of work (9-11 items) and compliance (12-13 items)]. SKAMP combined score is obtained by summing up each item score where each item is rated on a 7-point impairment scale (0=normal to 6=maximal impairment) for total possible combined score of 0 to 78; where higher score signified worst impairment. SKAMP deportment subscale is reported which assesses behavior in the classroom and comprises of 4 items, with a total possible score for each sub-scale of 0 to 24; higher score indicates worst impairment.
Time Frame: 0.75, 2, 4, 8, 10, 12 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NWP06 | Placebo
Number analyzed (Participants) | 39 | 39
units on a scale
  Hour 0.75 | 1.7 (1.89) | 3.3 (2.57)
  Hour 2 | 1.0 (1.39) | 3.6 (3.00)
  Hour 4 | 1.2 (1.64) | 4.2 (2.92)
  Hour 8 | 2.1 (3.03) | 4.5 (3.21)
  Hour 10 | 2.4 (2.98) | 3.7 (2.57)
  Hour 12 | 2.7 (2.91) | 4.2 (3.69)
Statistical Analysis 1: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean difference = -1.69, 95% CI 2-sided [-2.36 to -1.02], Standard Error of Mean 0.33
Statistical Analysis 2: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean difference = -2.66, 95% CI 2-sided [-3.50 to -1.82], Standard Error of Mean 0.41
Statistical Analysis 3: Comparison: NWP06 vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean difference = -2.95, 95% CI 2-sided [-3.77 to -2.13], Standard Error of Mean 0.40
Statistical Analysis 4: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean difference = -2.49, 95% CI 2-sided [-3.33 to -1.66], Standard Error of Mean 0.41
Statistical Analysis 5: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0035, ANOVA; LS mean difference = -1.26, 95% CI 2-sided [-2.07 to -0.44], Standard Error of Mean 0.40
Statistical Analysis 6: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.0109, ANOVA; LS mean difference = -1.43, 95% CI 2-sided [-2.51 to -0.35], Standard Error of Mean 0.53

5. Secondary Outcome: Permanent Product Measure of Performance (PERMP) Score Over 12 Hours
Description: The PERMP is a 10-minute written test, on 80 math problems, performed as seatwork in the classroom. At the end of the 10-minute math test , the PERMP score of the number of math problems attempted plus the number of math problems answered correctly in a 10-minute session was used to measure a participant's performance. The total score range from 0-160 with higher scores indicating better performance.
Time Frame: 0.75, 2, 4, 8, 10, 12 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NWP06 | Placebo
Number analyzed (Participants) | 39 | 39
units on a scale
  Hour 0.75 | 111.1 (62.40) | 85.5 (51.88)
  Hour 2 | 118.2 (63.87) | 82.4 (50.54)
  Hour 4 | 119.2 (64.31) | 75.5 (48.62)
  Hour 8 | 105.2 (63.94) | 72.1 (52.41)
  Hour 10 | 95.6 (63.64) | 82.7 (57.59)
  Hour 12 | 94.0 (61.69) | 78.1 (51.83)
Statistical Analysis 1: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean difference = 25.61, 95% CI 2-sided [16.26 to 34.96], Standard Error of Mean 4.61
Statistical Analysis 2: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean difference = 37.10, 95% CI 2-sided [26.54 to 47.66], Standard Error of Mean 5.21
Statistical Analysis 3: Comparison: NWP06 vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean difference = 45.77, 95% CI 2-sided [30.89 to 60.65], Standard Error of Mean 7.35
Statistical Analysis 4: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean difference = 35.46, 95% CI 2-sided [22.14 to 48.78], Standard Error of Mean 6.57
Statistical Analysis 5: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0155, ANOVA; LS mean difference = 14.86, 95% CI 2-sided [3.00 to 26.73], Standard Error of Mean 5.86
Statistical Analysis 6: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.0019, ANOVA; LS mean difference = 20.69, 95% CI 2-sided [8.17 to 33.22], Standard Error of Mean 6.18

6. Secondary Outcome: SKAMP Combined Scores Over 12 Hours
Description: The SKAMP scale measures the manifestations of attention deficit hyperactivity disorder (ADHD) using an independent observer rating of the participant's impairment in classroom observed behaviors. SKAMP combined score is comprised of 13 items (including subscales: attention with items 1-4, deportment with items 5-8, quality of work with items 9-11 and compliance with items 12-13). The SKAMP combined score was obtained by summing up each item score where each item is rated on a 7-point impairment scale (0=normal to 6=maximal impairment) for a total possible combined score of 0 to 78; where higher score signified worst impairment.
Time Frame: 0.75, 2, 8, 10, 12 hours post-dose
Population: Data for combined SKAMP score was collected and reported through the measure of onset and duration of clinical effects as given in outcome measure 2.
Groups:
- Placebo: Placebo-matched to NWP06 oral suspension once daily for 1 week in either of the 2 intervention period.
Arm/Group | NWP06 | Placebo
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: SKAMP Quality of Work Subscale Score Over 12 Hours
Description: SKAMP scale measures the manifestations of ADHD using an independent observer rating of the participant's impairment in classroom observed behaviors. SKAMP composite score is comprised of 13 items [subscales: attention (1-4 items), deportment (5-8 items), quality of work (9-11 items) and compliance (12-13 items)]. SKAMP composite score is obtained by summing up each item score where each item is rated on a 7-point impairment scale (0=normal to 6=maximal impairment) for total possible combined score of 0 to 78; where higher score signified worst impairment. SKAMP quality of work subscale is reported which comprises of 3 items, with a total possible score of 0 to 18; higher score indicates worst impairment.
Time Frame: 0.75, 2, 4, 8, 10, 12 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NWP06 | Placebo
Number analyzed (Participants) | 39 | 39
units on a scale
  Hour 0.75 | 4.6 (2.38) | 6.5 (3.06)
  Hour 2 | 3.8 (2.06) | 6.6 (3.03)
  Hour 4 | 3.6 (2.35) | 7.3 (3.34)
  Hour 8 | 5.5 (3.06) | 7.9 (3.19)
  Hour 10 | 6.4 (3.22) | 6.7 (2.71)
  Hour 12 | 6.5 (3.28) | 7.6 (3.66)
Statistical Analysis 1: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0014, ANOVA; LS mean difference = -1.80, 95% CI 2-sided [-2.85 to -0.74], Standard Error of Mean 0.52
Statistical Analysis 2: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean difference = -2.79, 95% CI 2-sided [-3.76 to -1.82], Standard Error of Mean 0.48
Statistical Analysis 3: Comparison: NWP06 vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean difference = -3.89, 95% CI 2-sided [-5.12 to -2.67], Standard Error of Mean 0.60
Statistical Analysis 4: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0002, ANOVA; LS mean difference = -2.65, 95% CI 2-sided [-3.97 to -1.33], Standard Error of Mean 0.65
Statistical Analysis 5: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.3492, ANOVA; LS mean difference = -0.43, 95% CI 2-sided [-1.34 to 0.49], Standard Error of Mean 0.45
Statistical Analysis 6: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.0105, ANOVA; LS mean difference = -1.34, 95% CI 2-sided [-2.34 to -0.33], Standard Error of Mean 0.50

8. Other Pre Specified Outcome: SKAMP Compliance Subscale Score Over 12 Hours
Description: SKAMP scale measures the manifestations of ADHD using an independent observer rating of the participant's impairment in classroom observed behaviors. SKAMP composite score is comprised of 13 items [subscales: attention (1-4 items), deportment (5-8 items), quality of work (9-11 items) and compliance (12-13 items)]. SKAMP composite score is obtained by summing up each item score where each item is rated on a 7-point impairment scale (0=normal to 6=maximal impairment) for total possible combined score of 0 to 78; where higher score signified worst impairment. SKAMP compliance subscale is reported which comprises of 2 items, with a total possible score of 0 to 12; higher score indicates worst impairment.
Time Frame: 0.75, 2, 4, 8, 10, 12 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NWP06 | Placebo
Number analyzed (Participants) | 39 | 39
units on a scale
  Hour 0.75 | 1.9 (1.96) | 3.5 (2.67)
  Hour 2 | 1.2 (1.51) | 4.1 (2.94)
  Hour 4 | 1.3 (1.77) | 4.7 (2.97)
  Hour 8 | 2.1 (2.46) | 4.8 (3.13)
  Hour 10 | 2.7 (3.01) | 4.4 (2.94)
  Hour 12 | 3.5 (3.16) | 4.6 (3.50)
Statistical Analysis 1: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean difference = -1.72, 95% CI 2-sided [-2.43 to -1.00], Standard Error of Mean 0.35
Statistical Analysis 2: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean difference = -2.94, 95% CI 2-sided [-3.78 to -2.10], Standard Error of Mean 0.41
Statistical Analysis 3: Comparison: NWP06 vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean difference = -3.34, 95% CI 2-sided [-4.11 to -2.57], Standard Error of Mean 0.38
Statistical Analysis 4: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean difference = -2.70, 95% CI 2-sided [-3.64 to -1.76], Standard Error of Mean 0.46
Statistical Analysis 5: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0006, ANOVA; LS mean difference = -1.57, 95% CI 2-sided [-2.40 to -0.73], Standard Error of Mean 0.41
Statistical Analysis 6: Comparison: NWP06 vs Placebo; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.0087, ANOVA; LS mean difference = -1.12, 95% CI 2-sided [-1.94 to -0.30], Standard Error of Mean 0.40

ADVERSE EVENTS:
Description: Safety population included all randomized participants who received at least 1 dose of study medication (either NWP06 or matching placebo) with at least 1 post-baseline safety assessment.
Groups:
- OL Phase (NWP06): NWP06 oral suspension once daily optimized during the 4 to 6 weeks open label phase at a starting dose of 20 milligram [mg] and titrated at a 10 or 20 mg increments, based on clinical response and tolerability to a maximum daily dose of 60 mg/day.
- DB Phase (Placebo): Placebo-matched to NWP06 oral suspension once daily for 1 week in either of the 2 intervention periods of the DB phase.
- DB Phase (NWP06): NWP06 oral suspension at a once daily optimized dose (optimized during the 4 to 6 weeks open label phase at a starting dose of 20 milligram [mg] and titrated at a 10 or 20 mg increments, based on clinical response and tolerability to a maximum daily dose of 60mg/day) for 1 week in either of the 2 intervention periods of the DB phase.
Arm/Group | OL Phase (NWP06) | DB Phase (Placebo) | DB Phase (NWP06)
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 42/45 | 5/45 | 11/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OL Phase (NWP06) (N=45) | DB Phase (Placebo) (N=45) | DB Phase (NWP06) (N=45)
Affect lability (Psychiatric disorders) | 12 | 1 | 4
Initial insomnia (Psychiatric disorders) | 10 | 0 | 1
Insomnia (Psychiatric disorders) | 8 | 0 | 0
Aggression (Psychiatric disorders) | 3 | 1 | 0
Logorrhoea (Psychiatric disorders) | 4 | 0 | 0
Change in sustained attention (Psychiatric disorders) | 2 | 0 | 0
Nail picking (Psychiatric disorders) | 2 | 0 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 | 0 | 0
Bruxism (Psychiatric disorders) | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Perseveration (Psychiatric disorders) | 0 | 0 | 1
Social avoidant behaviour (Psychiatric disorders) | 1 | 0 | 0
Stereotypy (Psychiatric disorders) | 0 | 1 | 0
Tic (Psychiatric disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 19 | 1 | 1
Vomiting (Gastrointestinal disorders) | 5 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 25 | 0 | 1
Headache (Nervous system disorders) | 8 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Mental impairment (Nervous system disorders) | 1 | 0 | 0
Oromandibular dystonia (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Sensory disturbance (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Irritability (General disorders) | 6 | 0 | 0
Fatigue (General disorders) | 4 | 0 | 0
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 2 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Viral rash (Infections and infestations) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Flushing (Vascular disorders) | 3 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 1 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Results for primary outcome is presented as absolute values and not as change from pre-dose and the secondary outcomes are presented at each post-dose time-point and not pre-dose, as planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.